CLINICAL TRIAL: NCT01222741
Title: Studies of Disorders With Increased Susceptibility to Fungal Infections
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100216; 10-I-0216
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-01

CONDITIONS: Fungal Infections; Primary Immune Deficiencies
Keywords: PID; Primary Immune Deficiencies; Candida; Immune Abnormalities; Diabetic; Natural History
MeSH Terms: conditions — Mycoses; Primary Immunodeficiency Diseases; Torulopsis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Voluntary: Healthy voluntary
- Patients: affected patient
- relatives: family member to patient

SUMMARY:
Background:

- Researchers are interested in studying disorders that make individuals more susceptible to fungal infections, specifically infections with the Candida yeast. These disorders are often related to problems with the immune system and may have genetic factors, which suggests that researchers should study not only the individual with the disorder, but also his or her first- and second-degree relatives (such as parents, siblings, children, and first cousins). To provide material for future research, individuals with immune disorders and their first- and second-degree relatives will be asked to provide blood and other samples for testing and comparison with samples taken from healthy volunteers with no history of immune disorders.

Objectives:

- To collect blood and other biological samples to study immune disorders that make individuals more susceptible to fungal infections.

Eligibility:

* Individuals of any age who have abnormal immune function characterized by recurrent or unusual fungal infections, recurrent or chronic inflammation, or other types of immune dysfunction.
* First- or second-degree genetically related family members (limited to mother, father, siblings, grandparents, children, aunts, uncles, and first cousins).
* Healthy volunteers at least 18 years of age (for comparison purposes).

Design:

* Participants will provide blood samples and buccal (cells from the inside of the mouth near the cheek) samples.
* Participants with immune disorders will also be asked to provide urine samples, saliva or mucosal samples, or skin tissue biopsies, and may also have imaging studies (such as x-rays) to collect information for research.
* Samples may be collected at the National Institutes of Health or at other clinical locations for the samples to the sent to the National Institutes of Health.
* No treatment will be provided as part of this protocol....

DETAILED DESCRIPTION:
This study is designed for the evaluation, diagnosis, and long-term follow up of selected patients with primary immune deficiencies and other conditions associated with fungal, and more specifically with Candida spp. infections. The primary immune deficiencies to be studied include, but are not limited to, autoimmune polyendocrinopathy candidiasis ectodermal dystrophy (APECED), chronic mucocutaneous candidiasis (CMC), myeloperoxidase deficiency (MPO), immune dysregulation polyendocrinopathy enteropathy X-linked (IPEX), Job s syndrome, chronic granulomatous disease (CGD), biotinidase deficiency, Ikaros zinc finger 1 (IKAROS)-associated diseases, and Interferon Regulatory Factor 4 (IRF4) deficiency. Diabetic patients and infants also show increased susceptibility to such infections and might be studied. Patient participants will undergo evaluations that include history/physical, blood sampling, genetic testing, and possible tissue sampling. We may use some of the blood cells to investigate the utility of induced pluripotent stem cells (iPS) for immune cell derivation and targeted gene correction. Relative participants who are first or second degree genetically related family members of patients (limited to mother, father, siblings, grandparents, children, aunts, uncles, and first cousins) might also be screened for clinical, in vitro, and genetic correlates of immune abnormalities. Healthy volunteers will be enrolled as a source of control samples for research testing. Among the aims of this protocol are to better understand the genetic and pathophysiologic factors that lead to defects in host defense, and to use modern and evolving methods in molecular and cellular biology to elucidate the pathogenesis of this particular susceptibility. A better understanding of primary immunodeficiency could allow for the rational development of novel therapies for such diseases and to benefit future patients, but it might not benefit current patient participants directly. Routine follow-up may occur every 6 months with evaluation and blood sampling. Under some circumstances, we may provide medically indicated standard treatments for the immune deficiencies under study, and we will collect information from clinically indicated care for research purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients

To be eligible to participate in this study as a patient, an individual must meet the following criteria:

* Be 2 years of age to be seen at the Clinical Center as an outpatient. Children <=3 years of age must not have severe infections, as assessed by the investigator, to be seen at the Clinical Center. Send-in samples may be submitted by participants >30 days of age.
* Have an abnormality of immune function as manifested by recurrent or unusual fungal infections, recurrent or chronic inflammation, or previous laboratory evidence of immune dysfunction. Of particular focus of this study are patients with:

  * APECED
  * CMC
  * MPO
  * IPEX
  * Hyper-immunoglobulin E syndrome (Job s syndrome)
  * CGD
  * Biotinidase deficiency
  * IKAROS defects
  * AIOLOS defects
  * IRF4 defects
  * Other conditions showing increased susceptibility to such infections as described in infants and type 1 diabetic patients
* Have a primary physician outside of the NIH.
* Agree to have blood stored for future research.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

Relatives

To be eligible to participate in this study as a relative, an individual must meet the following criteria:

* Be 2 years of age to be seen at the Clinical Center as an outpatient. Children <=3 years of age must not have severe infections, as assessed by the investigator, to be seen at the Clinical Center. Send-in samples may be submitted for participants >30 days of age.
* Be a mother, father, sibling, child, grandparent, aunt, uncle, or first cousin to a patient participant.
* Adult relatives must be able to provide informed consent.
* Agree to have blood stored for future research.

Healthy volunteers

To be eligible to participate in this study as a healthy volunteer, an individual must meet the following criteria:

* Be 18 to 85 years old.
* Have a hemoglobin count of >11 g/dL.
* Weigh >=110 pounds.
* Be able to provide informed consent.
* Be willing to have blood stored for future research.

EXCLUSION CRITERIA:

Patients and Relatives

In general, there are no strict exclusion criteria for these cohorts. However, the presence of certain types of acquired abnormalities of immunity solely due to HIV, chemotherapeutic agent(s), or an underlying malignancy could be grounds for possible exclusion for a patient or relative. In the opinion of the investigator, the presence of such disease processes may interfere with evaluation of a co-existing abnormality of immunity that is the subject of study under this protocol. Pregnant females will not be allowed to participate in any procedure that may be dangerous to the pregnancy or the fetus.

Healthy volunteers

An individual who meets any of the following criteria will be excluded from participation as a healthy volunteer in this study:

* Is receiving chemotherapeutic agent(s) or has an underlying malignancy.
* Is pregnant.
* Has a history of heart, lung, or kidney disease, or bleeding disorders.
* Has HIV or viral hepatitis (B or C), or history of viral hepatitis B or C since age 11.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with primary immune deficiencies, their first and second-degree blood relatives (relatives), and individuals with other conditions that result in increased susceptibility to Candida spp. infections. This study will also include healthy volunteer adults as a source of control samples.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2011-01-07 (Actual)

PRIMARY OUTCOMES:
characterization | 10 years
  Characterize and compare the clinical and laboratory features of APECED, CMC, and other primary immunodeficiencies or particular conditions (such as infancy or diabetic subjects) with increased susceptibility to Candida or other fungal infections.
Determine the prevalence of mutation | 10 years
  Determine the prevalence of AIRE mutations in patients with increased susceptibility to Candida or other fungal infections.
genotype-phenotype correlation | 10 years
  Establish a genotype-phenotype correlation in patients with different AIRE mutations.
Determine and compare the functionality | 10 years
  Determine and compare the functional integrity of Th17, Dectin1, and AIRE pathways in patients with increased susceptibility to Candida or other fungal infections with and without AIRE mutations

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Rosenzweig, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glocker EO, Hennigs A, Nabavi M, Schaffer AA, Woellner C, Salzer U, Pfeifer D, Veelken H, Warnatz K, Tahami F, Jamal S, Manguiat A, Rezaei N, Amirzargar AA, Plebani A, Hannesschlager N, Gross O, Ruland J, Grimbacher B. A homozygous CARD9 mutation in a family with susceptibility to fungal infections. N Engl J Med. 2009 Oct 29;361(18):1727-35. doi: 10.1056/NEJMoa0810719. PMID 19864672
- [Background] Plantinga TS, van der Velden WJ, Ferwerda B, van Spriel AB, Adema G, Feuth T, Donnelly JP, Brown GD, Kullberg BJ, Blijlevens NM, Netea MG. Early stop polymorphism in human DECTIN-1 is associated with increased candida colonization in hematopoietic stem cell transplant recipients. Clin Infect Dis. 2009 Sep 1;49(5):724-32. doi: 10.1086/604714. PMID 19614557
- [Background] Perheentupa J. Autoimmune polyendocrinopathy-candidiasis-ectodermal dystrophy. J Clin Endocrinol Metab. 2006 Aug;91(8):2843-50. doi: 10.1210/jc.2005-2611. Epub 2006 May 9. PMID 16684821
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0216.html